CLINICAL TRIAL: NCT00622596
Title: Prospective Cohort of Opiate Dependent Patients on Buprenorphine/Naloxone for Maintenance
Acronym: Project BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0504027630
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mobile Access to Buprenorphine (Experimental): High risk populations accessing a mobile health care system can obtain Buprenorphine for treatment.
  Interventions: Other: Mobile Access

INTERVENTIONS:
Other: Mobile Access — Subjects would access buprenorphine through mobile access. On day 1: 8 mg of buprenorphine, then on Day 2: 16 mg daily of buprenorphine sublingually.

SUMMARY:
The purpose of this study was to expand access to buprenorphine using a mobile health care system among marginalized populations with or at high risk for HIV and observe longitudinal effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV +
* At high risk for HIV (IV drug use, commercial sex worker, partner of HIV+)
* Mental Health (unmanaged or diagnosed mental illness)

Exclusion Criteria:

* Benzodiazepine use
* Opiate use due to pain management issues only (present or past)
* Non-IDU

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Attendance | 10/1/03-9/30/08
  To assess the feasibility and efficacy of the use of buprenorphine to treat opioid dependence in high risk populations accessing a mobile health care system using tracked attendance.
Opioid free urine toxicology | 10/1/03-9/30/08
  To assess the feasibility and efficacy of the use of buprenorphine to treat opioid dependence in high risk populations accessing a mobile health care system using incidence of opioid free urine toxicology.

SECONDARY OUTCOMES:
Access to other health care, incarceration, hospitalization acceptability of the site of care from both patient and provider perspectives, and attendance and adherence to counseling. | 10/1/03-9/30/08

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University School of Medicine/AIDS Program
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No